CLINICAL TRIAL: NCT01293136
Title: Retrospective Femoral Nerve Block Study
Status: Completed | Type: Observational
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Joseph D. Tobias, Chairman Dept. of Anesthesiology & Pain Medicine, Nationwide Children's Hospital
Other Study IDs: IRB11-00073
Record Dates: First submitted 2011-02-09; First posted 2011-02-10 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2012-01

CONDITIONS: Other Reconstructive Surgery
Keywords: knee; reconstructive surgery; femoral nerve block

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- intravenous opioids
  Interventions: Drug: Intravenous opioids
- femoral nerve block
  Interventions: Procedure: Femoral nerve block

INTERVENTIONS:
Procedure: Femoral nerve block — Ropivacaine
  Groups: femoral nerve block
Drug: Intravenous opioids — Whatever opioids prescribed
  Groups: intravenous opioids

SUMMARY:
This is a retrospective review to evaluate the efficacy of femoral nerve block in providing analgesia following reconstructive surgery of the knee and to compare the postoperative course of patients who received femoral nerve block with a retrospective cohort who were cared for prior to the institution of a regional anesthesia program. The investigators hypothesize that femoral nerve blockade limits postoperative opioid needs, improves analgesia and facilitates discharge home when compared to intravenous opioid use following reconstructive knee surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients that had reconstructive knee surgery between July 2009 to the present.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients that had reconstructive knee surgery
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2011-02; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Duration of hospitalization | 1 Week
  duration of hospitalization and need for inpatient admission in patients who received femoral nerve block versus those who received intravenous opioids

SECONDARY OUTCOMES:
Nausea and vomiting | 1 Week
Total opioid use | 1 Week
Postoperative pain score | 1 Week

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States